CLINICAL TRIAL: NCT02463890
Title: Effect of Exercise Training on Obstructive Sleep Apnea Syndrome Severity
Acronym: EXESAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1508033; 2015-A00490-49 (Other: ANSM)
Record Dates: First submitted 2015-06-03; First posted 2015-06-04 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Sleep Apnea Syndromes; Sleep Apnea, Obstructives
Keywords: Sleep Apnea Syndromes; Sleep Apnea, Obstructives; Training
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): In this group, patients will perform 3 sessions of one hour per week of the "NeuroGyV" training program. It is a physical activity program with one session of Nordic walking, one session of "aquagym" and one session of gymnastic. Program lasts 9 months.
  Interventions: Other: Training
- Control (Other): In this group, patients will receive only diets and physical activity counselling
  Interventions: Other: Control

INTERVENTIONS:
Other: Training
  Other Names: NeuroGyV program
  Arms: Training
Other: Control
  Arms: Control

SUMMARY:
Sleep apnoea affects more than 20% of people over 65 years and is largely underdiagnosed. It does multiply tenfold the occurrence of vascular events, particularly stroke. While Continuous Positive Airway Pressure (CPAP) is currently the Gold standard treatment to prevent cerebrovascular and cardiovascular events, with a major clinical benefit, long term adherence to CPAP is a significant problem and search for alternative treatment is essential.

The investigators hypothesize that long-term exercise training would allow to reduce significantly sleep apnoea syndrome severity. Thus, in this study, the investigators will compare evolution of Apnoea Hypopnea Index (AHI) in an exercise trained group performed through in a national based non-profit organization (Fédération Française d'éducation Physique et de Gymnastique Volontaire (FFEPGV)) using a medical established program (NeuroGyV) during nine months against a control group receiving only standard dietetic and physical activity counseling.

ELIGIBILITY:
Inclusion Criteria:

* Patients affiliated or entitled to a social security system
* Patients with AHI from 15 to 30 per hour
* Signature of consent

Exclusion Criteria:

* Patients being already treated for sleep apnea or clinical status (cardiovascular comorbidities) justifying an immediate initiation of CPAP
* Daytime sleepiness (ESS score > 10)
* Known respiratory or heart disease (or discovering during stress test) contraindicated exercise training
* Patients with Parkinson's disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Final polysomnography | 9 months
  Percentage of patients with AHI < 15/hour through polysomnography assessment after nine months of follow-up in the training and the control groups

SECONDARY OUTCOMES:
First intermediate polysomnography | 3 months
  Percentage of patients with AHI<15/hour through polysomnography assessment after three months of follow-up in the training and the control groups.
Second intermediate polysomnography | 6 months
  Percentage of patients with AHI<15/hour through polysomnography assessment after six months of follow-up in the training and the control groups.
High frequency | 9 months
  Correlation between change in AHI and change in high frequency (HF) of spectral analysis of heart rate variability (parasympathetic index) at 9 months of follow-up in the 2 groups
Maximal aerobic capacity (VO2Max) | 9 months
  Correlation between the change in VO2max during stress test, walking distance during 6 minutes and AHI in the two groups
Population Physical Activity questionnaire (POPAQ) | 9 months
  Correlation between the change in daily physical activity energy expenditure (estimated by the POPAQ questionnaire) and AHI in the two groups
Daily physical activity energy expenditure | 9 months
  Correlation between the daily physical activity energy expenditure (estimated directly by an actimetry sensor for 7 days) and AHI in the two groups
Epworth sleepiness Scale | 9 months
  Comparison of the variation of Epworth Sleepiness Scale (ESS) after 9 months follow-up for the two groups
Pittsburgh questionnaire | 9 months
  Comparison of the variation of Pittsburgh questionnaire after 9 months follow-up for the two groups
Berlin questionnaire | 9 months
  Comparison of the variation of Berlin questionnaire after 9 months follow-up for the two groups
Blood pressure - Baroreflex | 9 months
  Measure of autonomic function (parasympathetic activity) - quantified via changes in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ROCHE, MD - PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger M, Barthelemy JC, Hupin D, Raffin J, Dupre C, Labeix P, Costes F, Gaspoz JM, Roche F. Benefits of supervised community physical activity in obstructive sleep apnoea. Eur Respir J. 2018 Nov 22;52(5):1801592. doi: 10.1183/13993003.01592-2018. Print 2018 Nov. No abstract available. PMID 30361248
- See also: Website of the FFEPGV (in french) — http://www.sport-sante.fr/accueil/